CLINICAL TRIAL: NCT06951256
Title: Dexmedetomidine as an Adjuvant to Bupivacaine in Scalp Block Versus Bupivacaine Alone for Intraoperative Mean Arterial Pressure Stability in Adult Patients Undergoing Craniotomy
Brief Title: Dexmedetomidine as an Adjuvant to Bupivacaine in Scalp Block vs Bupivacaine Alone for Hemodynamics Stability in Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS78/2024
Record Dates: First submitted 2025-04-04; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-03

CONDITIONS: Dexmedetomidine; Craniotomy; Regional Anesthesia; Mean Arterial Pressure Stability
Keywords: Scalp block; Mean arterial pressure stability; Dexmedetomidine; Craniotomy
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group SB (n =18 patient) will receive scalp block with Bupivacaine alone. (Active Comparator): In Group SB: 20 ml of Bupivacaine 0.25% was given Scalp nerve block was done under complete aseptic condition where local infiltration of local anesthetic (LA) was done guided by bony superficial landmarks to block the supraorbital, supratrochlear, auriculotemporal, occipital, and post auricular branches of the greater auricular nerves.
  In both group maximal dose of Bupivacaine was not exceed (2.5 mg/kg).
  Interventions: Drug: Scalp block with bupivacaine alone
- Group SD (n =18 patient) will receive scalp block with dexmedetomidine as an adjuvant to Bupivacaine (Active Comparator): In group SD: local infiltration of total volume 20 ml which include (Bupivacaine 0.25%. + Dexmedetomidine 1 mcg/kg) was given.
  Dexmedetomidine preparation was done by 2 ml (200 mcg) diluted by 18 ml normal saline in 20 ml syringe as 1 ml was contained 10 mcg and was used.
  Scalp block was given by the same way as group SB. In both group maximal dose of Bupivacaine was not exceed (2.5 mg/kg).
  Interventions: Drug: Scalp block by adding dexmedetomidine as an adjuvant to bupivacaine

INTERVENTIONS:
Drug: Scalp block with bupivacaine alone — In Group SB: (LA) was done by 20ml of Bupivacaine 0.25%. maximal dose of Bupivacaine did not exceed (2.5 mg/kg) Scalp nerve block will be done by anesthesiologist who is blind to the drug being injected and under complete septic condition where local infiltration of local anesthetic (LA) will be done guided by bony superficial landmarks to block the supraorbital, supratrochlear, auriculotemporal, occipital, and post auricular branches of the greater auricular nerves
  Other Names: Traditional scalp block
  Arms: Group SB (n =18 patient) will receive scalp block with Bupivacaine alone.
Drug: Scalp block by adding dexmedetomidine as an adjuvant to bupivacaine — local infiltration of total volume 20ml which include (Bupivacaine 0.25%. + Dexmedetomidine 1mcg/kg) was done Dexmedetomidine preparation was done by 2ml (200 mcg) diluted by 18 ml normal saline in 20 ml syringe as 1ml was contain 10 mcg and injected at same points as above
  Other Names: Scalp block by dexmedetomidine; Dexmedetomidine; Dexmedetomidine as an adjuvant to bupivacaine
  Arms: Group SD (n =18 patient) will receive scalp block with dexmedetomidine as an adjuvant to Bupivacaine

SUMMARY:
The investigator tested the effect of dexmedetomidine as an adjuvant to bupivacaine compared to bupivacaine alone in mean arterial pressure stability in adult patients undergoing craniotomy

DETAILED DESCRIPTION:
A) Preoperative settings:

Complete history taking and full physical examination. Routine preoperative investigations was done to all patients including laboratory investigations (complete blood picture, liver function tests, prothrombin time and partial thromboplastin time) and other as needed by the patient condition.

Written informed consent was obtained from all participants prior to the study. Patients was educated visual analogue score for pain (VAS), which consisted of 10c.m line, with two end points (where 0=no pain and 10=worst pain).

B) Intraoperative settings:

Electrocardiogram (ECG), non-invasive blood pressure (NIBP), pulse oximeter (SpO2) will be applied, and baseline readings were taken before induction, no sedation was given.

Anesthesia was induced after a period of preoxygenation with 100% oxygen for 2-3 minutes with intravenous injection of fentanyl 2 µg/kg .propofol 2 mg/kg ) and a muscle relaxant (Atracurium) 0.5 mg/kg after loss of patient consciousness.

After endotracheal intubation, intubation was confirmed by ETCO2 and bilateral auscultation of the chest.

Anesthesia was maintained with 60% oxygen mixed with air and isoflurane 1-2%. Lungs were ventilated using volume-controlled ventilation with tidal volumes and respiratory rate adjusted to maintain end tidal CO2 at 35-40 mmHg.

Following anesthesia induction, a continuous invasive blood pressure monitoring was initiated through radial 20-gauge arterial catheterization, as well as urine output through bladder catheterization.

Sampling method:

The patients were randomly divided into two equal groups using a computerized generated list (closed opaque sealed envelope).

Group SB (n =18 patient) received scalp block with Bupivacaine alone. Group SD (n =18 patient) received scalp block with Dexmedetomidine as an adjuvant to Bupivacaine.

In both group:

Scalp nerve block was done by anesthesiologist who is blind to the drug being injected and under complete septic condition where local infiltration of local anesthetic (LA) was done guided by bony superficial landmarks to block the supraorbital, supratrochlear, auriculotemporal, occipital, and post auricular branches of the greater auricular nerves as follow :

The patient lied supine on the table while the performing operator usually stands at the head end facing the feet.

The supraorbital and supratrochlear nerves were blocked with 2 mL of solution as they emerge from the orbit with needle introduced above the eyebrow perpendicular to the skin. The supraorbital notch was located by palpation, and the needle was introduced perpendicularly 1 cm medial to the notch.

The auriculotemporal nerves was performed with the patient's head turned to one side so that the side to be blocked faces upward with 3 mL of solution injected 1.5 cm anterior to the ear at the level of the tragus; the needle was introduced perpendicular to the skin and infiltration made deep to the fascia and superficially as the needle withdrawn. The superficial temporal artery should be palpated to avoid intra-arterial injection. Negative aspiration is a must for this block.

The post auricular branches of the greater auricular nerves were blocked with 2 mL of solution between skin and bone, 1.5 cm posterior to the ear at the level of the tragus The needle was inserted at 90 degrees till bony contact is made, upon which it is withdrawn, and subcutaneous injection was performed.

The greater, lesser, and third occipital nerves were blocked with 3 mL of solution with infiltration along the superior nuchal line, approximately halfway between the occipital protuberance and the mastoid process.

In Group SB: (LA) was done by 20ml of Bupivacaine 0.25%.

While Group SD:

local infiltration of total volume 20ml which include (Bupivacaine 0.25%. + Dexmedetomidine 1mcg/kg) was done.

In both group maximal dose of Bupivacaine didn't not exceed (2.5 mg/kg) . Dexmedetomidine preparation was done by 2ml (200 mcg) diluted by 18 ml normal saline in 20 ml syringe as 1ml was contain 10 mcg and used.

Mayfield placement in all patients was done 15 minutes after scalp block was given.

*Both blocks was done & or supervised by an expert all through. At the end of the surgery, the residual neuromuscular block was be reversed with intravenous injection of neostigmine (0.05 mg/kg) with atropine (0.01 mg/kg), Endotracheal tube extubation was done and then the patient was transferred to Postoperative anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 65 years.
* Patients ASA I or II undergoing supratentorial elective planned craniotomies.

Exclusion Criteria:

* Patients refused to participate in the study.
* Patients with cardiovascular diseases such as hypertension or low cardiac reserve.
* History or known allergy to the used local anesthetic or opioids.
* Patient could not understand a visual analog scale (VAS).
* Bleeding disorders.
* Evidence of local infection at site of injection. 7. Emergency craniotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative mean arterial pressure measured after Mayfeild insertion during craniotomies. | During the operation
  Mean blood pressure (MAP) was monitored continuously and recorded at Base line, before Mayfield placement, after 5mins of Mayfield insertion and at the end of surgery. The hemodynamic parameters at each step of recording were compared between the two groups.

SECONDARY OUTCOMES:
Surgeon satisfaction as regard surgical field. Postoperative VAS score and time for 1st rescue analgesia. Total analgesic consumption in first 24 hours postoperative. | During 24 hours
  1. Heart rate was monitored continuously and recorded at Base line, before Mayfield placement, after 5mins of Mayfield insertion and at the end of surgery. The hemodynamic parameters at each step of recording were compared between the two groups.
  2. Intraoperative surgeon satisfaction:
     Surgeon satisfaction regard surgical field was assessed and recorded according to a 5-point Likert scale (5: excellent, 4: Good, 3: Satisfactory, 2: Poor, 1: Very poor).
  3. Assessment of post-operative pain:
  Post operatively, the patient was transferred to the PACU where pain intensity was evaluated on a (0-10) visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Yara Sa Ghareb, MBBCH, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After paper publication
Supporting Information: Study Protocol, SAP, ICF